CLINICAL TRIAL: NCT06961630
Title: A Pilot Randomized Trial of Post-Operative Biomarker-Guided Precision Medicine With Rivaroxaban and Atorvastatin for Cardiovascular Risk-Reduction
Brief Title: Post-Operative Biomarker-Guided Precision Medicine For Cardiovascular Risk Reduction
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-01260; 1R34HL173301-01A1 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Injury After Noncardiac Surgery
MeSH Terms: interventions — Rivaroxaban; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rivaroxaban + Atorvastatin (Experimental): Participants assigned to this arm will receive rivaroxaban 2.5mg twice daily + atorvastatin 80mg daily for 6 months.
  Interventions: Drug: Rivaroxaban; Drug: Atorvastatin
- Usual Care (No Intervention): Participants assigned to usual care will continue all clinically indicated therapies as prescribed by their treating physicians.

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 2.5mg will be orally administered twice daily for 6 months.
  Arms: Rivaroxaban + Atorvastatin
Drug: Atorvastatin — Atorvastatin 80mg will be orally administered daily for 6 months.
  Arms: Rivaroxaban + Atorvastatin

SUMMARY:
The goal of this pilot study is to assess enrollment feasibility of a randomized trial of direct oral anticoagulant and high-intensity statin therapy versus usual care in patients with Myocardial Injury after Noncardiac Surgery (MINS). The primary aims of this study are to assess feasibility, study drug adherence, and optimize study design (entry criteria, study endpoints, sample size calculation, site selection) and recruitment strategies for the future multicenter randomized clinical trial studying biomarker-based care in post-operative patients at elevated cardiovascular (CV) risk.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥45 years
2. Underwent major non-cardiac surgery requiring ≥1 overnight inpatient stay in the prior 14 days
3. Myocardial injury after noncardiac surgery, defined as a post-operative troponin ≥ 99th percentile upper reference limit [URL], with rise/fall >20% indicative of acute myocardial injury.
4. Ability to provide informed consent

Exclusion Criteria:

1. Expected survival <6 months
2. Hemorrhagic disorder
3. Surgeon feels it is unsafe to initiate low-dose anticoagulation within 14 days of surgery
4. Indication for oral anticoagulation at discharge
5. Indication for dual antiplatelet therapy at discharge
6. Patient already receiving or planned to receive moderate or high-intensity statin
7. Contraindication to high-intensity statin
8. Contraindication to rivaroxaban
9. End stage kidney disease on hemodialysis
10. Acute liver failure or decompensated cirrhosis
11. Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of pills taken at Month 6 | Month 6
  Treatment adherence will be assessed by pill count and patient self report.

SECONDARY OUTCOMES:
Percentage of Quality of Life (QOL) questionnaires completed at Month 6 | Month 6
  Two QOL questionnaires (Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS-10) and EuroQol 5 Dimension (EQ5D)) will be administered at baseline, 2-month follow-up visit, and the 6-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel R. Smilowitz, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared for any purpose immediately following publication. No end date. Data are available indefinitely at: NHLBI BioData Catalyst (BDC), an existing NIH-supported Scientific Data Repository. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Data are available indefinitely for anyone who wishes to access the data for any purpose at: NHLBI BioData Catalyst (BDC), an existing NIH-supported Scientific Data Repository.
URL: https://biodatacatalyst.nhlbi.nih.gov/